CLINICAL TRIAL: NCT04884100
Title: enHEART - Exploring Full Content of Optical Signals to Enhance Cardiac Arrhythmia Screening
Acronym: enHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Prof. Etienne Pruvot, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-00586
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Atrioventricular Block; Nodal Tachycardia; Atrioventricular Tachycardia; Ventricular Tachycardia; Premature Ventricular Contraction; Premature Atrial Complex
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Atrioventricular Block; Tachycardia, Ventricular; Ventricular Premature Complexes; Atrial Premature Complexes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PPG recording (Other): arrhythmia recording using PPG monitor
  Interventions: Other: Validating and improving PPG-based algorithms

INTERVENTIONS:
Other: Validating and improving PPG-based algorithms — Our project aims at validating and improving PPG-based algorithms that were previously developed during the time course of a preceding study mini-Holter, accepted by the CER-VD in 2015. The developed features might help improve our understanding of the physio-pathological expression of cardiac arrhythmias. Indeed, current evidence demonstrates that PPG signals contain rich information on diverse cardiovascular mechanisms and properties

SUMMARY:
This research will investigate the PPG signal morphology related to physiological and non- physiological changes in arrhythmia-related heart rate as well as the performance of the PPG-based features previously developed within the framework of the Mini-Holter study to discriminate between several cardiac arrhythmias. To this end, clinical data will be recorded on patients by using a wrist-based PPG monitor simultaneously with 12-lead ECG and intracardiac electrogram (EGM) signals at the university hospital in Lausanne. Importantly, this study will remain purely observational as it will not change the diagnostic and therapeutic management of the included patients, nor will it interfere with the time course of the procedures. The aim of enHEART study is to validate on a larger database the ability of several previously developed PPG-based features to detect a variety of cardiac arrhythmias.

DETAILED DESCRIPTION:
The aim of the study is to acquire high quality PPG signals of various types of cardiac arrhythmias during diagnostic and therapeutic procedures, under controlled conditions (i.e., electrophysiology lab), which can be compared beat-to-beat to a concurrently-acquired, gold-standard reference (12-lead ECG and intracardiac EGM signals), and expert annotations by CHUV physicians. To this end, a total of 99 patients referred for diagnostic or therapeutic interventions (ablation) of 9 different types of cardiac arrhythmias at the CHUV will be enrolled. 11 patients per type of arrhythmia will be included.

The following clinical data will be collected from the electronic file of the patient:

1. Clinical data such as age, gender, weight, size, BMI, blood pressure and heart rate, cardiovascular risk factors, clinical history
2. Baseline treatment and treatment at time of the electrophysiological procedure
3. Arrhythmia type and arrhythmia-related symptoms
4. Left and right ventricular ejection fraction as provided by the patient's private cardiologist echocardiogram.

The following paraclinical data will be synchronously collected during the diagnostic and/or therapeutic intervention in the electrophysiology laboratory:

1. Surface ECG signals
2. Intracardiac EGM signals as provided by the intracardiac catheters used for the diagnostic and/or therapeutic interventions. Depending on the type of intervention, up to three different catheters may be used
3. PPG signals as provided by the PPG wrist monitor

The primary objective of our study is to investigate if features extracted from the pulse morphology of PPG signals (waveform-based features) significantly improve the classification accuracy of cardiac arrhythmias compared to a classification based on heart rate variation (HRV) features only.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18-year-old,
2. Able to speak/read/understand French,
3. Informed consent signed, and
4. at least one of the following cardiac arrhythmias:

   * sustained or non-sustained ventricular tachycardia,
   * sustained or non-sustained atrial tachycardia
   * atrial flutter,
   * frequent atrial and/or ventricular ectopic beats,
   * ventricular and/or atrial bigeminy,
   * left bundle branch block,
   * second- or third-degree atrioventricular block,
   * atrioventricular reentrant tachycardia or atrioventricular node reentrant tachycardia,
   * AF

Exclusion Criteria:

1. Patient is pregnant or breastfeeding,
2. Refusal of participation by the patient
3. Patient is less than 18 years old,
4. Patient incapable of judgement or under tutelage, or
5. Patient is already included in another human research project (ClinO/HRO) that may affect the objectives of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Performances of cardiac arrhythmias classification based on Photoplethysmography (PPG) signals. | 2 years
  Standard statistical quantities related to a classification task will be reported: accuracy, sensitivity, specificity, positive predictive value, F1 score and area under the receiver operating characteristics curve.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne PRUVOT, Professor, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland